CLINICAL TRIAL: NCT04298580
Title: Randomized, Single-Blinded Study to Evaluate the Timing Effect of Ultrasound-Guided Paravertebral Block in Patients Undergoing Robotic Mitral Valve Repair Procedure
Brief Title: Timing Effect of Ultrasound-Guided PVB After Robotic Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Manxu Zhao, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000203
Record Dates: First submitted 2020-02-25; First posted 2020-03-06 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Nerve Block; Cardiac Surgery
Keywords: Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVB before surgery (Active Comparator)
  Interventions: Procedure: PVB block
- PVB after surgery (Active Comparator)
  Interventions: Procedure: PVB block

INTERVENTIONS:
Procedure: PVB block — PVB block before surgery versus after surgery

SUMMARY:
This study is to evaluate whether the administration of ultrasound-guided paravertebral block (PVB) after surgery would produce better postoperative pain control and fast postoperative recovery after Robotic cardiac surgery. Half of participants will receive PVB before surgery, while the other half will receive PVB at the end of surgery.

DETAILED DESCRIPTION:
Ultrasound-guided PVB (either before surgery, or after surgery) is the standard postoperative pain management for Robotic cardiac surgery. This technique is to inject local anesthetic (numb medication) around nerve to decrease pain. But the optimal time of PVB is unknown.

The administration of PVB before surgery can help pain control during the surgery and after surgery. But the duration of PVB could be reduced because surgery itself can last 5-6 hrs.

The PVB after surgery will not provide pain control during surgery, but may provide longer pain control after surgery, and may help participants faster recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 yrs
2. ASA I-IV
3. Either gender

Exclusion Criteria:

1. Refusal to participate in the study
2. Age< 18 yrs
3. Contraindications to regional blockage including but not limited to:

   1. Patient refusal to regional blockade
   2. Infection at the site of needle insertion
   3. Systemic infection
   4. Bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Durations of ICU and hospitalization | 2-6 days
  Duration (days) of ICU stay, and duration of hospital stay

SECONDARY OUTCOMES:
Pain intensity measure | 2-3 days
  self reported pain intensity at every 4 hour while in the ICU. It is a scored 0-10 (0 = no pain, 10 + pain as bad as can be)

IPD SHARING:
Plan to Share IPD: No